CLINICAL TRIAL: NCT02752841
Title: The Effect of Vitamin D Repletion on Urinary Calcium Excretion in Kidney Stone Formers With Vitamin D Deficiency and High Urinary Calcium
Brief Title: The Effect of Vitamin D Repletion on Kidney Stone Risk
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited study funding
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Jie Tang, Associate Professor, Brown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 879658-1
Record Dates: First submitted 2016-04-20; First posted 2016-04-27 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Calculi
MeSH Terms: conditions — Calculi | interventions — Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Nutritional vitamin D repletion and maintenance
  Interventions: Dietary Supplement: Nutritional vitamin D repletion and maintenance

INTERVENTIONS:
Dietary Supplement: Nutritional vitamin D repletion and maintenance — Ergocalciferol (50,000 IU weekly for 12 weeks) for vitamin D repletion, ergocalciferol (50,000 IU monthly) or cholecalciferol (1000 IU daily) for maintenance of vitamin D

SUMMARY:
Examine the effect of nutritional vitamin D repletion on urinary calcium excretion and kidney stone burden in calcium kidney stone formers

DETAILED DESCRIPTION:
The investigators plan to conduct a clinic-based interventional study of 50 patients followed at Miriam Hospital Kidney Stone Clinic with history of nephrolithiasis, urinary calcium excretion between 150 and 400 mg/day, and 25-vitamin D deficiency/insufficiency (defined as serum level ≤ 30ng/ml). The intervention is oral ergocalciferol 50,000 IU per week for 12 weeks (repletion course). After that, the same repletion course will be repeated if serum 25-vitamin D remains ≤ 30ng/ml or drops to ≤ 30ng/ml anytime during the study. Otherwise, a maintenance dose of cholecalciferol 1,000 IU daily or ergocalciferol 50,000 IU monthly will be prescribed for the rest of the study. Each participant will serve as his own control. The outcome is the change in urinary calcium excretion and stone burden assessed by renal ultrasound. The planned study duration is 12 months. The investigators will have greater than 95% power to detect a 10% increase in 24-hour urinary calcium.

ELIGIBILITY:
Inclusion Criteria:

* History of nephrolithiasis
* 25(OH)D deficiency (defined as serum level ≤ 30ng/ml) within 3 months of enrollment
* 24-hour urinary calcium excretion > 150 mg/day and < 400 mg/day (measured less than 2 months prior to study enrollment)

Exclusion Criteria:

* Known uric acid, cystine, or struvite stone disease
* Hypercalcemia (serum calcium >10.4 mg/dl within the past 12 months)
* Gross hematuria within the past 6 months
* Acute stone event within the past 1 month
* Recent stone intervention within the past 1 month
* Suspected or known secondary causes of hypercalciuria such as primary hyperparathyroidism, sarcoidosis, hyperthyroidism, or malignancy (except non-melanoma skin cancer)
* Addition or dose change of medicines potentially affecting urinary calcium since enrollment 24-hour urine collection (including diuretics, magnesium supplements, potassium supplements, potassium citrate, and vitamin D supplementation)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in urinary calcium excretion measured by timed urine collection | Baseline and 12 months
  Examine changes in urine calcium excretion at the end of the 12month study. Urinary calcium excretion are measured by 24-hour urine collections for calcium (mg per day), and the differences are the changes of 24-hour urine calcium (mg per day) between those measured at month 12 and at the enrollment

SECONDARY OUTCOMES:
Changes in kidney stone burden measured by ultrasound | Baseline and 12 months
  Changes in kidney stone burden at the end of the 12month study. Total stone burden is calculated by number of stones x stone sizes, i.e., patient A has one stone measured at 2 mm and two stones measured at 3 mm, then total stone burden = 1x2 +2x3=8mm.

IPD SHARING:
Plan to Share IPD: Undecided